CLINICAL TRIAL: NCT01342211
Title: A Phase 2, Double-blind, Placebo-controlled, Randomized Study To Assess The Efficacy, Safety And Tolerability Of Pf-04950615 Following Multiple Intravenous Doses In Hypercholesterolemic Subjects On High Doses Of Atorvastatin, Rosuvastatin Or Simvastatin.
Brief Title: A Multiple Dose Study of PF-04950615 (RN316) in Subjects on High Doses of Statins
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: B1481005
Record Dates: First submitted 2011-04-25; First posted 2011-04-27 (Estimated); Results first posted 2017-10-11 (Actual); Last update posted 2017-10-11 (Actual); Status verified 2017-09

CONDITIONS: Hypercholesterolemia; Dyslipidemia
Keywords: PF-04950615; RN316
MeSH Terms: conditions — Hypercholesterolemia; Dyslipidemias | interventions — Hydroxymethylglutaryl-CoA Reductase Inhibitors; bococizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Treatment A (Placebo Comparator)
  Interventions: Biological: Placebo; Drug: Statin
- Treatment B (Experimental)
  Interventions: Biological: PF-04950615 (RN316); Drug: Statin
- Treatment C (Experimental)
  Interventions: Biological: PF-04950615 (RN316); Drug: Statin
- Treatment D (Experimental)
  Interventions: Biological: PF-04950615 (RN316); Drug: Satin
- Treatment E (Experimental)
  Interventions: Biological: PF-04950615 (RN316); Drug: Statin

INTERVENTIONS:
Biological: Placebo — Intravenous placebo monthly during treatment phase.
  Arms: Treatment A
Drug: Statin — Single daily dose of atorvastatin (40 or 80 mg), rosuvastatin (20 or 40 mg) or simvastatin (40 or 80 mg) from Day 1 to Day 141/ET.
  Arms: Treatment A
Biological: PF-04950615 (RN316) — Intravenous 10mg/mL based on weight monthly during treatment phase.
  Arms: Treatment B
Drug: Statin — Single daily dose of atorvastatin (40 or 80 mg), rosuvastatin (20 or 40 mg) or simvastatin (40 or 80 mg) from Day 1 to Day 141/ET.
  Arms: Treatment B
Biological: PF-04950615 (RN316) — Intravenous 10mg/mL based on weight monthly during treatment phase.
  Arms: Treatment C
Drug: Statin — Single daily dose of atorvastatin (40 or 80 mg), rosuvastatin (20 or 40 mg) or simvastatin (40 or 80 mg) from Day 1 to Day 141/ET.
  Arms: Treatment C
Biological: PF-04950615 (RN316) — Intravenous 10mg/mL based on weight monthly during treatment phase.
  Arms: Treatment D
Drug: Satin — Single daily dose of atorvastatin (40 or 80 mg), rosuvastatin (20 or 40 mg) or simvastatin (40 or 80 mg) from Day 1 to Day 141/ET.
  Arms: Treatment D
Biological: PF-04950615 (RN316) — Intravenous 10mg/mL based on weight monthly during treatment phase.
  Arms: Treatment E
Drug: Statin — Single daily dose of atorvastatin (40 or 80 mg), rosuvastatin (20 or 40 mg) or simvastatin (40 or 80 mg) from Day 1 to Day 141/ET.
  Arms: Treatment E

SUMMARY:
This study will investigate the effect of PF-04950615, a new investigational lipid lowering agent, on LDL-C and other lipids.

ELIGIBILITY:
Inclusion Criteria:

* On a stable daily dose of atorvastatin, rosuvastatin or simvastatin.
* Lipids meet the following criteria at screening and prior to dosing: Fasting LDL-C greater than 100 mg/dL and fasting TG less than 400 mg/dL

Exclusion Criteria:

* History of a cardiovascular or cerebrovascular event or procedure during the past year.
* Poorly controlled type 1 or type 2 diabetes mellitus.
* Poorly controlled hypertension.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2011-07 (Actual); Primary Completion 2012-02 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (44):
- United States (38):
  - Orange County Research Center, Tustin, California
  - Diablo Clinical Research, Inc., Walnut Creek, California
  - Innovative Research of West Florida, Inc., Clearwater, Florida
  - Avail Clinical Research, LLC, DeLand, Florida
  - In Vivo Clinical Research, Inc., Doral, Florida
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - Kendall South Medical Center, Miami, Florida
  - North Georgia Clinical Research, Woodstock, Georgia
  - North Georgia Internal Medicine, Woodstock, Georgia
  - Vince and Associates Clinical Research, Overland Park, Kansas
  - Heartland Research Associates, LLC, Wichita, Kansas
  - L-MARC Research Center, Louisville, Kentucky
  - Commonwealth Biomedical Research, LLC, Madisonville, Kentucky
  - Maine Research Associates, Auburn, Maine
  - Infinity Medical Research, North Dartmouth, Massachusetts
  - Saint Luke's Hospital, Kansas City, Missouri
  - Saint Luke's Lipid and Diabetes Research Center, Kansas City, Missouri
  - The Center for Pharmaceutical Research, P.C., Kansas City, Missouri
  - Medex Healthcare Research, Inc., St Louis, Missouri
  - New Mexico Clinical Research & Osteoporosis Center, Incorporated, Albuquerque, New Mexico
  - North Carolina Clinical Research, Raleigh, North Carolina
  - PMG Research of Salisbury, Salisbury, North Carolina
  - Lynn Health Science Institute, Oklahoma City, Oklahoma
  - Oklahoma Cardiovascular Research Group (OCRG), Oklahoma City, Oklahoma
  - Oklahoma Heart Hospital Physicians, Oklahoma City, Oklahoma
  - Oklahoma Heart Hospital, Oklahoma City, Oklahoma
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - Perelman Center for Advanced Medicine, Philadelphia, Pennsylvania
  - Translational Research Center, Philadelphia, Pennsylvania
  - Spartanburg Medical Research, Spartanburg, South Carolina
  - New Orleans Center for Clinical Research, Knoxville, Tennessee
  - Volunteer Research Group, Knoxville, Tennessee
  - Texas Center for Drug Development, Inc., Houston, Texas
  - Paragon Research Center, LLC, San Antonio, Texas
  - Clinical Trials of Texas, Inc., San Antonio, Texas
  - San Antonio Preventive & Diagnostic Medicine, PA, San Antonio, Texas
  - National Clinical Research - Norfolk, Inc., Norfolk, Virginia
  - National Clinical Research - Richmond, Inc., Richmond, Virginia
- Canada (6):
  - The Medical Arts Health Research Group, Kelowna, British Columbia
  - Q & T Research Chicoutimi, Chicoutimi, Quebec
  - Centre de Recherche Clinique de Laval, Laval, Quebec
  - Diex Research Montreal Inc., Montreal, Quebec
  - Clinique des Maladies Lipidiques de Quebec Inc., Québec, Quebec
  - Diex Research Sherbrooke Inc., Sherbrooke, Quebec

REFERENCES:
- [Derived] Wang EQ, Kaila N, Plowchalk D, Gibiansky L, Yunis C, Sweeney K. Population PK/PD modeling of low-density lipoprotein cholesterol response in hypercholesterolemic participants following administration of bococizumab, a potent anti-PCSK9 monoclonal antibody. CPT Pharmacometrics Syst Pharmacol. 2023 Dec;12(12):2013-2026. doi: 10.1002/psp4.13050. Epub 2023 Nov 22. PMID 37994400
- [Derived] Wan H, Gumbiner B, Joh T, Riel T, Udata C, Forgues P, Garzone PD. Effects of Proprotein Convertase Subtilisin/Kexin Type 9 (PCSK9) Inhibition with Bococizumab on Lipoprotein Particles in Hypercholesterolemic Subjects. Clin Ther. 2017 Nov;39(11):2243-2259.e5. doi: 10.1016/j.clinthera.2017.09.009. Epub 2017 Oct 14. PMID 29037448
- [Derived] Udata C, Garzone PD, Gumbiner B, Joh T, Liang H, Liao KH, Williams JH, Meng X. A Mechanism-Based Pharmacokinetic/Pharmacodynamic Model for Bococizumab, a Humanized Monoclonal Antibody Against Proprotein Convertase Subtilisin/Kexin Type 9, and Its Application in Early Clinical Development. J Clin Pharmacol. 2017 Jul;57(7):855-864. doi: 10.1002/jcph.867. Epub 2017 Feb 9. PMID 28181260
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1481005&StudyName=A%20Multiple%20Dose%20Study%20of%20PF-04950615%20%28RN316%29%20in%20Subjects%20on%20High%20Doses%20of%20Statins

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Participants received intravenous infusion of placebo (normal saline) on Day 1, 29 and 57 along with atorvastatin or simvastatin (40 or 80 milligram [mg]) or rosuvastatin (20 or 40 mg) tablet orally once daily from Day 1 to 141.
- PF-04950615 0.25 mg/kg: Participants received intravenous infusion of PF-04950615 (RN316) 0.25 milligram per kilogram (mg/kg) on Day 1, 29 and 57 along with atorvastatin or simvastatin (40 or 80 mg) or rosuvastatin (20 or 40 mg) tablet orally once daily from Day 1 to 141.
- PF-04950615 1.0 mg/kg: Participants received intravenous infusion of PF-04950615 (RN316) 1.0 mg/kg on Day 1, 29 and 57 along with atorvastatin or simvastatin (40 or 80 mg) or rosuvastatin (20 or 40 mg) tablet orally once daily from Day 1 to 141.
- PF-04950615 3.0 mg/kg: Participants received intravenous infusion of PF-04950615 (RN316) 3.0 mg/kg on Day 1, 29 and 57 along with atorvastatin or simvastatin (40 or 80 mg) or rosuvastatin (20 or 40 mg) tablet orally once daily from Day 1 to 141.
- PF-04950615 6.0 mg/kg: Participants received intravenous infusion of PF-04950615 (RN316) 6.0 mg/kg on Day 1, 29 and 57 along with atorvastatin or simvastatin (40 or 80 mg) or rosuvastatin (20 or 40 mg) tablet orally once daily from Day 1 to 141.
Period: Overall Study
Arm/Group | Placebo | PF-04950615 0.25 mg/kg | PF-04950615 1.0 mg/kg | PF-04950615 3.0 mg/kg | PF-04950615 6.0 mg/kg
Started | 19 | 19 | 18 | 19 | 18
Treated | 19 | 17 | 18 | 19 | 17
Completed | 19 | 17 | 18 | 17 | 16
Not Completed | 0 | 2 | 0 | 2 | 2
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 0
Not completed — Randomized, but not Treated | 0 | 2 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety analysis population included all participants who received at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | PF-04950615 0.25 mg/kg | PF-04950615 1.0 mg/kg | PF-04950615 3.0 mg/kg | PF-04950615 6.0 mg/kg | Total
Number analyzed (Participants) | 19 | 17 | 18 | 19 | 17 | 90
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.2 (12.4) | 57.9 (10.3) | 56.3 (9.1) | 58.0 (10.6) | 60.8 (5.7) | 58.4 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 9 | 11 | 11 | 8 | 45
  Male | 13 | 8 | 7 | 8 | 9 | 45

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Low-density Lipoprotein Cholesterol (LDL-C) at Day 85
Description: Baseline value was calculated as the average of Day 7 and Day 1 measurements collected prior to study drug administration.
Time Frame: Baseline, Day 85
Population: Efficacy analysis set included all participants who received at least 1 dose of study drug and completed the Day 85 visit or dropped out prematurely, whichever was earlier. Here 'N' (Overall number of participants analyzed) signifies participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | PF-04950615 0.25 mg/kg | PF-04950615 1.0 mg/kg | PF-04950615 3.0 mg/kg | PF-04950615 6.0 mg/kg
Number analyzed (Participants) | 18 | 16 | 18 | 18 | 17
percent change | -8.91 (20.075) | -13.11 (20.786) | -8.63 (30.394) | -47.20 (31.021) | -56.48 (35.289)
Statistical Analysis 1: Comparison: Placebo vs PF-04950615 0.25 mg/kg; Analysis was performed using analysis of covariance (ANCOVA) model with fixed effects for treatment, background statin, treatment by background statin interaction, and baseline; Test type: Superiority or Other; p = 0.5661, ANCOVA; Least squares (LS) Mean Difference = -5.63, 95% CI 2-sided [-25.09 to 13.83], Standard Error of Mean 9.759
Statistical Analysis 2: Comparison: Placebo vs PF-04950615 1.0 mg/kg; Analysis was performed using ANCOVA model with fixed effects for treatment, background statin, treatment by background statin interaction, and baseline; Test type: Superiority or Other; p = 0.8080, ANCOVA; LS Mean Difference = -2.30, 95% CI 2-sided [-21.08 to 16.49], Standard Error of Mean 9.422
Statistical Analysis 3: Comparison: Placebo vs PF-04950615 3.0 mg/kg; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.0001, ANCOVA; LS Mean Difference = -37.72, 95% CI 2-sided [-56.47 to -18.97], Standard Error of Mean 9.404
Statistical Analysis 4: Comparison: Placebo vs PF-04950615 6.0 mg/kg; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p < 0.0001, ANCOVA; LS Mean Difference = -49.11, 95% CI 2-sided [-68.08 to -30.14], Standard Error of Mean 9.514

2. Secondary Outcome: Percentage of Participants Achieving Low-density Lipoprotein Cholesterol (LDL-C) Less Than (<) 70 and <100 Milligram Per Deciliter (mg/dL)
Time Frame: Day 29, 57, 85
Population: Efficacy analysis set included all participants who received at least 1 dose of study drug and completed the Day 85 visit or dropped out prematurely, whichever was earlier. 'N' = participants who were evaluable for this outcome measure and 'number analyzed' = participants who were evaluable at specified time points for each arm.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | PF-04950615 0.25 mg/kg | PF-04950615 1.0 mg/kg | PF-04950615 3.0 mg/kg | PF-04950615 6.0 mg/kg
Number analyzed (Participants) | 19 | 16 | 18 | 18 | 17
percentage of participants
  Day 29 <70 mg/dL: number analyzed (Participants) | 19 | 16 | 17 | 18 | 16
  Day 29 <70 mg/dL | 5.3 | 6.3 | 11.8 | 77.8 | 100
  Day 29 <100 mg/dL: number analyzed (Participants) | 19 | 16 | 17 | 18 | 16
  Day 29 <100 mg/dL | 47.4 | 18.8 | 35.3 | 94.4 | 100
  Day 57 <70 mg/dL: number analyzed (Participants) | 17 | 15 | 15 | 18 | 17
  Day 57 <70 mg/dL | 0 | 0 | 0 | 44.4 | 76.5
  Day 57 <100 mg/dL: number analyzed (Participants) | 17 | 15 | 15 | 18 | 17
  Day 57 <100 mg/dL | 47.1 | 13.3 | 53.3 | 66.7 | 88.2
  Day 85 <70 mg/dL: number analyzed (Participants) | 18 | 16 | 18 | 18 | 17
  Day 85 <70 mg/dL | 5.6 | 0 | 11.1 | 66.7 | 64.7
  Day 85 <100 mg/dL: number analyzed (Participants) | 18 | 16 | 18 | 18 | 17
  Day 85 <100 mg/dL | 33.3 | 50.0 | 33.3 | 88.9 | 76.5
Statistical Analysis 1: Comparison: Placebo vs PF-04950615 0.25 mg/kg; Day 29, <70 mg/dL: The standard logistic regression model was used to assess treatment effect; Test type: Superiority or Other; p = 0.8998, Regression, Logistic; Odds Ratio (OR) = 1.172, 95% CI 2-sided [0.10 to 13.92]
Statistical Analysis 2: Comparison: Placebo vs PF-04950615 1.0 mg/kg; Day 29, <70 mg/dL: The standard logistic regression model was used to assess treatment effect; Test type: Superiority or Other; p = 0.5273, Regression, Logistic; Odds Ratio (OR) = 2.063, 95% CI 2-sided [0.22 to 19.48]
Statistical Analysis 3: Comparison: Placebo vs PF-04950615 3.0 mg/kg; Day 29, <70 mg/dL: The standard logistic regression model was used to assess treatment effect; Test type: Superiority or Other; p = 0.0004, Regression, Logistic; Odds Ratio (OR) = 53.924, 95% CI 2-sided [5.93 to 490.67]
Statistical Analysis 4: Comparison: Placebo vs PF-04950615 6.0 mg/kg; Day 29, <70 mg/dL: The standard logistic regression model was used to assess treatment effect; Test type: Superiority or Other; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 280.366, 95% CI 2-sided [18.65 to 4214.35]
Statistical Analysis 5: Comparison: Placebo vs PF-04950615 0.25 mg/kg; Day 29, <100 mg/dL: The standard logistic regression model was used to assess treatment effect; Test type: Superiority or Other; p = 0.0860, Regression, Logistic; Odds Ratio (OR) = 0.262, 95% CI 2-sided [0.06 to 1.21]
Statistical Analysis 6: Comparison: Placebo vs PF-04950615 1.0 mg/kg; Day 29, <100 mg/dL: The standard logistic regression model was used to assess treatment effect; Test type: Superiority or Other; p = 0.4308, Regression, Logistic; Odds Ratio (OR) = 0.579, 95% CI 2-sided [0.15 to 2.25]
Statistical Analysis 7: Comparison: Placebo vs PF-04950615 3.0 mg/kg; Day 29, <100 mg/dL: The standard logistic regression model was used to assess treatment effect; Test type: Superiority or Other; p = 0.0127, Regression, Logistic; Odds Ratio (OR) = 8.272, 95% CI 2-sided [1.57 to 43.56]
Statistical Analysis 8: Comparison: Placebo vs PF-04950615 6.0 mg/kg; Day 29, <100 mg/dL: The standard logistic regression model was used to assess treatment effect; Test type: Superiority or Other; p = 0.0096, Regression, Logistic; Odds Ratio (OR) = 13.528, 95% CI 2-sided [1.89 to 97.00]
Statistical Analysis 9: Comparison: Placebo vs PF-04950615 0.25 mg/kg; Day 57, <70 mg/dL: The standard logistic regression model was used to assess treatment effect; Test type: Superiority or Other; p = 0.9519, Regression, Logistic; Odds Ratio (OR) = 1.131, 95% CI 2-sided [0.02 to 61.54]
Statistical Analysis 10: Comparison: Placebo vs PF-04950615 1.0 mg/kg; Day 57, <70 mg/dL: The standard logistic regression model was used to assess treatment effect; Test type: Superiority or Other; p = 0.9740, Regression, Logistic; Odds Ratio (OR) = 1.069, 95% CI 2-sided [0.02 to 58.00]
Statistical Analysis 11: Comparison: Placebo vs PF-04950615 3.0 mg/kg; Day 57, <70 mg/dL: The standard logistic regression model was used to assess treatment effect; Test type: Superiority or Other; p = 0.0273, Regression, Logistic; Odds Ratio (OR) = 28.286, 95% CI 2-sided [1.46 to 549.78]
Statistical Analysis 12: Comparison: Placebo vs PF-04950615 6.0 mg/kg; Day 57, <70 mg/dL: The standard logistic regression model was used to assess treatment effect; Test type: Superiority or Other; p = 0.0022, Regression, Logistic; Odds Ratio (OR) = 114.508, 95% CI 2-sided [5.50 to 2384.03]
Statistical Analysis 13: Comparison: Placebo vs PF-04950615 0.25 mg/kg; Day 57, <100 mg/dL: The standard logistic regression model was used to assess treatment effect; Test type: Superiority or Other; p = 0.0684, Regression, Logistic; Odds Ratio (OR) = 0.216, 95% CI 2-sided [0.04 to 1.12]
Statistical Analysis 14: Comparison: Placebo vs PF-04950615 1.0 mg/kg; Day 57, <100 mg/dL: The standard logistic regression model was used to assess treatment effect; Test type: Superiority or Other; p = 0.9068, Regression, Logistic; Odds Ratio (OR) = 1.081, 95% CI 2-sided [0.29 to 3.99]
Statistical Analysis 15: Comparison: Placebo vs PF-04950615 3.0 mg/kg; Day 57, <100 mg/dL: The standard logistic regression model was used to assess treatment effect; Test type: Superiority or Other; p = 0.2235, Regression, Logistic; Odds Ratio (OR) = 2.251, 95% CI 2-sided [0.61 to 8.31]
Statistical Analysis 16: Comparison: Placebo vs PF-04950615 6.0 mg/kg; Day 57, <100 mg/dL: The standard logistic regression model was used to assess treatment effect; Test type: Superiority or Other; p = 0.0120, Regression, Logistic; Odds Ratio (OR) = 8.250, 95% CI 2-sided [1.59 to 42.82]
Statistical Analysis 17: Comparison: Placebo vs PF-04950615 0.25 mg/kg; Day 85, <70 mg/dL: The standard logistic regression model was used to assess treatment effect; Test type: Superiority or Other; p = 0.5449, Regression, Logistic; Odds Ratio (OR) = 0.359, 95% CI 2-sided [0.01 to 9.92]
Statistical Analysis 18: Comparison: Placebo vs PF-04950615 1.0 mg/kg; Day 85, <70 mg/dL: The standard logistic regression model was used to assess treatment effect; Test type: Superiority or Other; p = 0.5585, Regression, Logistic; Odds Ratio (OR) = 1.914, 95% CI 2-sided [0.22 to 16.85]
Statistical Analysis 19: Comparison: Placebo vs PF-04950615 3.0 mg/kg; Day 85, <70 mg/dL: The standard logistic regression model was used to assess treatment effect; Test type: Superiority or Other; p = 0.0022, Regression, Logistic; Odds Ratio (OR) = 21.059, 95% CI 2-sided [3.00 to 147.65]
Statistical Analysis 20: Comparison: Placebo vs PF-04950615 6.0 mg/kg; Day 85, <70 mg/dL: The standard logistic regression model was used to assess treatment effect; Test type: Superiority or Other; p = 0.0020, Regression, Logistic; Odds Ratio (OR) = 22.851, 95% CI 2-sided [3.15 to 165.99]
Statistical Analysis 21: Comparison: Placebo vs PF-04950615 0.25 mg/kg; Day 85, <100 mg/dL: The standard logistic regression model was used to assess treatment effect; Test type: Superiority or Other; p = 0.3750, Regression, Logistic; Odds Ratio (OR) = 1.844, 95% CI 2-sided [0.48 to 7.12]
Statistical Analysis 22: Comparison: Placebo vs PF-04950615 1.0 mg/kg; Day 85, <100 mg/dL: The standard logistic regression model was used to assess treatment effect; Test type: Superiority or Other; p = 0.9140, Regression, Logistic; Odds Ratio (OR) = 1.078, 95% CI 2-sided [0.28 to 4.23]
Statistical Analysis 23: Comparison: Placebo vs PF-04950615 3.0 mg/kg; Day 85, <100 mg/dL: The standard logistic regression model was used to assess treatment effect; Test type: Superiority or Other; p = 0.0036, Regression, Logistic; Odds Ratio (OR) = 9.548, 95% CI 2-sided [2.09 to 43.57]
Statistical Analysis 24: Comparison: Placebo vs PF-04950615 6.0 mg/kg; Day 85, <100 mg/dL: The standard logistic regression model was used to assess treatment effect; Test type: Superiority or Other; p = 0.0149, Regression, Logistic; Odds Ratio (OR) = 6.093, 95% CI 2-sided [1.42 to 26.10]

3. Secondary Outcome: Percentage of Participants Achieving at Least 30 Percent Decrease in Low-density Lipoprotein Cholesterol (LDL-C)
Time Frame: Day 29, 57, 85
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | PF-04950615 0.25 mg/kg | PF-04950615 1.0 mg/kg | PF-04950615 3.0 mg/kg | PF-04950615 6.0 mg/kg
Number analyzed (Participants) | 19 | 16 | 18 | 18 | 17
percentage of participants
  Day 29: number analyzed (Participants) | 19 | 16 | 17 | 18 | 16
  Day 29 | 15.8 | 25.0 | 11.8 | 88.9 | 100
  Day 57: number analyzed (Participants) | 17 | 15 | 15 | 18 | 17
  Day 57 | 11.8 | 0 | 26.7 | 55.6 | 76.5
  Day 85: number analyzed (Participants) | 18 | 16 | 18 | 18 | 17
  Day 85 | 16.7 | 18.8 | 22.2 | 66.7 | 82.4
Statistical Analysis 1: Comparison: Placebo vs PF-04950615 0.25 mg/kg; Day 29: The standard logistic regression model was used to assess treatment effect; Test type: Superiority or Other; p = 0.5436, Regression, Logistic; Odds Ratio (OR) = 1.674, 95% CI 2-sided [0.32 to 8.83]
Statistical Analysis 2: Comparison: Placebo vs PF-04950615 1.0 mg/kg; Day 29: The standard logistic regression model was used to assess treatment effect; Test type: Superiority or Other; p = 0.7420, Regression, Logistic; Odds Ratio (OR) = 0.734, 95% CI 2-sided [0.12 to 4.63]
Statistical Analysis 3: Comparison: Placebo vs PF-04950615 3.0 mg/kg; Day 29: The standard logistic regression model was used to assess treatment effect; Test type: Superiority or Other; p = 0.0002, Regression, Logistic; Odds Ratio (OR) = 28.151, 95% CI 2-sided [4.73 to 167.62]
Statistical Analysis 4: Comparison: Placebo vs PF-04950615 6.0 mg/kg; Day 29: The standard logistic regression model was used to assess treatment effect; Test type: Superiority or Other; p = 0.0001, Regression, Logistic; Odds Ratio (OR) = 71.214, 95% CI 2-sided [7.88 to 643.42]
Statistical Analysis 5: Comparison: Placebo vs PF-04950615 0.25 mg/kg; Day 57: The standard logistic regression model was used to assess treatment effect; Test type: Superiority or Other; p = 0.3210, Regression, Logistic; Odds Ratio (OR) = 0.203, 95% CI 2-sided [0.01 to 4.74]
Statistical Analysis 6: Comparison: Placebo vs PF-04950615 1.0 mg/kg; Day 57: The standard logistic regression model was used to assess treatment effect; Test type: Superiority or Other; p = 0.3786, Regression, Logistic; Odds Ratio (OR) = 2.175, 95% CI 2-sided [0.39 to 12.27]
Statistical Analysis 7: Comparison: Placebo vs PF-04950615 3.0 mg/kg; Day 57: The standard logistic regression model was used to assess treatment effect; Test type: Superiority or Other; p = 0.0144, Regression, Logistic; Odds Ratio (OR) = 7.576, 95% CI 2-sided [1.50 to 38.38]
Statistical Analysis 8: Comparison: Placebo vs PF-04950615 6.0 mg/kg; Day 57: The standard logistic regression model was used to assess treatment effect; Test type: Superiority or Other; p = 0.0007, Regression, Logistic; Odds Ratio (OR) = 20.465, 95% CI 2-sided [3.59 to 116.60]
Statistical Analysis 9: Comparison: Placebo vs PF-04950615 0.25 mg/kg; Day 85: The standard logistic regression model was used to assess treatment effect; Test type: Superiority or Other; p = 0.8626, Regression, Logistic; Odds Ratio (OR) = 1.161, 95% CI 2-sided [0.21 to 6.30]
Statistical Analysis 10: Comparison: Placebo vs PF-04950615 1.0 mg/kg; Day 85: The standard logistic regression model was used to assess treatment effect; Test type: Superiority or Other; p = 0.6237, Regression, Logistic; Odds Ratio (OR) = 1.497, 95% CI 2-sided [0.30 to 7.51]
Statistical Analysis 11: Comparison: Placebo vs PF-04950615 3.0 mg/kg; Day 85: The standard logistic regression model was used to assess treatment effect; Test type: Superiority or Other; p = 0.0072, Regression, Logistic; Odds Ratio (OR) = 8.029, 95% CI 2-sided [1.76 to 36.65]
Statistical Analysis 12: Comparison: Placebo vs PF-04950615 6.0 mg/kg; Day 85: The standard logistic regression model was used to assess treatment effect; Test type: Superiority or Other; p = 0.0005, Regression, Logistic; Odds Ratio (OR) = 20.557, 95% CI 2-sided [3.73 to 113.20]

4. Secondary Outcome: Change From Baseline in Lipid Parameters at Day 29, 57 and 85
Description: Lipid parameters included: high-density lipoprotein cholesterol (HDL-C), total cholesterol (TC), non-high-density lipoprotein-cholesterol (non-HDL-C), triglyceride (TG), apolipoprotein B (ApoB) and apolipoprotein A1 (ApoA1). Baseline value was calculated as the average of Day 7 and Day 1 measurements collected prior to study drug administration.
Time Frame: Baseline, Day 29, 57, 85
Population: Efficacy analysis set. 'number analyzed' = participants who were evaluable at specified time points for each arm. Results for change at Day 85 in lipid parameters ApoB and ApoA1 were not reported because data was not collected for ApoB and ApoA1 at Day 85 due to an inadvertent omission in the protocol.
Measure: Mean (Standard Deviation); unit: milligram per deciliter (mg/dL)
Arm/Group | Placebo | PF-04950615 0.25 mg/kg | PF-04950615 1.0 mg/kg | PF-04950615 3.0 mg/kg | PF-04950615 6.0 mg/kg
Number analyzed (Participants) | 19 | 17 | 18 | 19 | 17
milligram per deciliter (mg/dL)
  Baseline: HDL-C | 46.18 (10.235) | 51.53 (14.084) | 49.11 (13.291) | 50.24 (11.724) | 44.76 (8.189)
  Baseline: TC | 202.82 (27.96) | 202.03 (27.10) | 205.11 (22.64) | 202.66 (37.98) | 206.91 (35.96)
  Baseline: Non-HDL-C | 156.63 (30.61) | 150.50 (29.03) | 156.00 (24.08) | 152.42 (38.89) | 162.15 (37.82)
  Baseline: TG | 136.18 (58.82) | 137.62 (87.56) | 162.83 (85.68) | 118.05 (47.08) | 172.47 (86.49)
  Baseline: ApoB | 106.74 (19.86) | 105.76 (18.21) | 109.83 (23.61) | 102.84 (22.06) | 109.06 (29.49)
  Baseline: ApoA1 | 140.32 (21.71) | 153.76 (22.73) | 146.44 (20.35) | 143.11 (20.31) | 141.29 (16.25)
  Change at Day 29: HDL-C: number analyzed (Participants) | 19 | 16 | 17 | 18 | 17
  Change at Day 29: HDL-C | 0.87 (5.627) | 3.59 (7.265) | 0.79 (5.041) | 4.50 (4.624) | 6.00 (6.072)
  Change at Day 29:TC: number analyzed (Participants) | 19 | 16 | 17 | 18 | 17
  Change at Day 29:TC | -10.66 (31.13) | -9.97 (29.104) | -21.94 (15.93) | -81.00 (49.61) | -111.68 (28.7)
  Change at Day 29: Non-HDL-C: number analyzed (Participants) | 19 | 16 | 17 | 18 | 17
  Change at Day 29: Non-HDL-C | -11.53 (33.16) | -13.56 (28.17) | -22.74 (14.91) | -85.50 (48.59) | -117.68 (25.9)
  Change at Day 29: TG: number analyzed (Participants) | 19 | 16 | 17 | 18 | 17
  Change at Day 29: TG | 8.66 (46.865) | -3.72 (31.384) | -37.03 (66.12) | -18.97 (48.88) | -46.94 (65.20)
  Change at Day 29: ApoB: number analyzed (Participants) | 19 | 16 | 17 | 18 | 14
  Change at Day 29: ApoB | -5.05 (16.119) | -9.56 (18.155) | -13.24 (15.63) | -47.13 (23.85) | -67.40 (22.03)
  Change at Day 29: ApoA1: number analyzed (Participants) | 19 | 16 | 17 | 18 | 14
  Change at Day 29: ApoA1 | 1.68 (10.546) | 2.06 (17.117) | 4.29 (11.751) | 11.67 (14.892) | 7.29 (12.875)
  Change at Day 57: HDL-C: number analyzed (Participants) | 17 | 15 | 15 | 18 | 17
  Change at Day 57: HDL-C | -0.74 (5.310) | 2.23 (8.113) | 2.83 (8.004) | 3.17 (7.462) | 4.88 (7.167)
  Change at Day 57: TC: number analyzed (Participants) | 17 | 15 | 15 | 18 | 17
  Change at Day 57: TC | -13.97 (28.37) | -5.67 (18.777) | -8.20 (39.052) | -51.33 (52.08) | -79.21 (52.81)
  Change at Day 57: Non-HDL-C: number analyzed (Participants) | 17 | 15 | 15 | 18 | 17
  Change at Day 57: Non-HDL-C | -13.24 (29.52) | -7.90 (21.123) | -11.03 (39.49) | -54.50 (55.71) | -84.09 (54.92)
  Change at Day 57: TG: number analyzed (Participants) | 17 | 15 | 15 | 18 | 17
  Change at Day 57: TG | -1.24 (61.405) | -11.37 (36.99) | -15.73 (95.34) | -4.47 (74.402) | -26.71 (49.54)
  Change at Day 57: ApoB: number analyzed (Participants) | 17 | 15 | 15 | 18 | 17
  Change at Day 57: ApoB | -8.94 (14.355) | -1.07 (12.384) | -3.87 (27.302) | -29.07 (31.83) | -45.90 (36.60)
  Change at Day 57: ApoA1: number analyzed (Participants) | 17 | 15 | 15 | 18 | 17
  Change at Day 57: ApoA1 | -2.59 (15.500) | -0.13 (14.020) | 8.47 (18.917) | 8.39 (20.448) | 10.12 (14.168)
  Change at Day 85: HDL-C: number analyzed (Participants) | 18 | 16 | 18 | 18 | 17
  Change at Day 85: HDL-C | 0.08 (5.219) | 1.81 (9.377) | 1.44 (5.739) | 5.50 (7.310) | 4.82 (7.671)
  Change at Day 85: TC: number analyzed (Participants) | 18 | 16 | 18 | 18 | 17
  Change at Day 85: TC | -10.97 (24.41) | -20.56 (31.99) | -11.56 (43.45) | -62.89 (52.73) | -79.97 (55.39)
  Change at Day 85: Non-HDL-C: number analyzed (Participants) | 18 | 16 | 18 | 18 | 17
  Change at Day 85: Non-HDL-C | -11.06 (26.14) | -22.38 (34.45) | -13.00 (40.28) | -68.39 (54.01) | -84.79 (52.95)
  Change at Day 85: TG: number analyzed (Participants) | 18 | 16 | 18 | 18 | 17
  Change at Day 85: TG | 2.97 (59.087) | -25.97 (49.96) | -9.39 (63.159) | -6.58 (58.104) | -40.12 (73.83)

5. Secondary Outcome: Percent Change From Baseline in Lipid Parameters at Day 29, 57 and 85
Description: as for outcome 4
Time Frame: Baseline, Day 29, 57, 85
Population: Efficacy analysis set. 'number analyzed' = participants who were evaluable at specified time points for each arm. Results for percent change at Day 85 for ApoB and ApoA1 were not reported because data was not collected for ApoB and ApoA1 at Day 85 due to an inadvertent omission in the protocol.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | PF-04950615 0.25 mg/kg | PF-04950615 1.0 mg/kg | PF-04950615 3.0 mg/kg | PF-04950615 6.0 mg/kg
Number analyzed (Participants) | 19 | 17 | 18 | 19 | 17
percent change
  Percent change at Day 29: HDL-C: number analyzed (Participants) | 19 | 16 | 17 | 18 | 17
  Percent change at Day 29: HDL-C | 1.98 (11.164) | 5.88 (12.764) | 0.27 (9.020) | 9.34 (10.291) | 12.96 (12.116)
  Percent change at Day 29: TC: number analyzed (Participants) | 19 | 16 | 17 | 18 | 17
  Percent change at Day 29: TC | -5.03 (15.148) | -3.88 (14.148) | -10.62 (7.813) | -38.54 (19.844) | -53.52 (7.450)
  Percent change at Day 29:Non-HDL-C: number analyzed (Participants) | 19 | 16 | 17 | 18 | 17
  Percent change at Day 29:Non-HDL-C | -7.14 (20.758) | -7.57 (17.933) | -14.75 (10.320) | -54.06 (23.588) | -73.23 (9.029)
  Percent change at Day 29: TG: number analyzed (Participants) | 19 | 16 | 17 | 18 | 17
  Percent change at Day 29: TG | 9.83 (35.146) | -0.50 (26.358) | -15.79 (27.131) | -15.94 (34.219) | -22.55 (31.973)
  Percent change at Day 29: ApoB: number analyzed (Participants) | 19 | 16 | 17 | 18 | 14
  Percent change at Day 29: ApoB | -4.09 (14.429) | -7.67 (15.315) | -11.27 (14.177) | -44.93 (18.320) | -61.17 (9.142)
  Percent change at Day 29: ApoA1: number analyzed (Participants) | 19 | 16 | 17 | 18 | 14
  Percent change at Day 29: ApoA1 | 1.24 (7.493) | 1.50 (10.896) | 2.88 (7.949) | 8.75 (11.114) | 5.55 (9.613)
  Percent change at Day 57: HDL-C: number analyzed (Participants) | 17 | 15 | 15 | 18 | 17
  Percent change at Day 57: HDL-C | -1.09 (10.708) | 4.96 (17.618) | 6.01 (15.077) | 6.78 (15.755) | 11.06 (15.390)
  Percent change at Day 57: TC: number analyzed (Participants) | 17 | 15 | 15 | 18 | 17
  Percent change at Day 57: TC | -6.91 (13.742) | -2.27 (8.829) | -3.85 (18.857) | -24.17 (22.496) | -37.36 (21.167)
  Percent change at Day 57: Non-HDL-C: number analyzed (Participants) | 17 | 15 | 15 | 18 | 17
  Percent change at Day 57: Non-HDL-C | -8.34 (18.789) | -4.26 (12.999) | -6.97 (23.977) | -34.84 (31.588) | -50.78 (26.254)
  Percent change at Day 57: TG: number analyzed (Participants) | 17 | 15 | 15 | 18 | 17
  Percent change at Day 57: TG | 5.90 (42.384) | -2.62 (21.430) | 1.66 (53.893) | -5.70 (53.271) | -10.76 (32.710)
  Percent change at Day 57: ApoB: number analyzed (Participants) | 17 | 15 | 15 | 18 | 17
  Percent change at Day 57: ApoB | -8.32 (13.214) | -0.61 (12.068) | -1.51 (23.582) | -27.25 (28.265) | -40.06 (29.448)
  Percent change at Day 57: ApoA1: number analyzed (Participants) | 17 | 15 | 15 | 18 | 17
  Percent change at Day 57: ApoA1 | -1.70 (11.575) | 0.57 (9.918) | 5.31 (11.150) | 6.81 (15.094) | 7.81 (12.152)
  Percent change at Day 85: HDL-C: number analyzed (Participants) | 18 | 16 | 18 | 18 | 17
  Percent change at Day 85: HDL-C | 0.87 (10.121) | 3.58 (19.489) | 3.00 (12.481) | 10.67 (13.967) | 10.70 (17.738)
  Percent change at Day 85: TC: number analyzed (Participants) | 18 | 16 | 18 | 18 | 17
  Percent change at Day 85: TC | -5.44 (12.468) | -9.45 (14.947) | -5.52 (20.658) | -28.78 (22.023) | -36.55 (26.150)
  Percent change at Day 85: Non-HDL-C: number analyzed (Participants) | 18 | 16 | 18 | 18 | 17
  Percent change at Day 85: Non-HDL-C | -6.78 (17.417) | -13.11 (20.428) | -8.48 (24.291) | -41.28 (27.815) | -50.16 (32.255)
  Percent change at Day 85: TG: number analyzed (Participants) | 18 | 16 | 18 | 18 | 17
  Percent change at Day 85: TG | 6.16 (42.923) | -8.14 (37.105) | -1.90 (37.939) | -4.22 (42.180) | -14.11 (40.324)

6. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. Serious adverse event (SAE) was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. TEAEs are events between first dose of study drug and up to Day 141 that were absent before treatment or that worsened relative to pretreatment state. Treatment related: a TEAE deemed related to the study drug by the investigator. TEAEs included SAEs (TESAEs) as well as non-serious AEs which occurred during the study. The participants with TEAEs, SAEs and treatment-related TEAEs were reported.
Time Frame: Day 1 up to Day 141
Population: Safety analysis set included all participants who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | Placebo | PF-04950615 0.25 mg/kg | PF-04950615 1.0 mg/kg | PF-04950615 3.0 mg/kg | PF-04950615 6.0 mg/kg
Number analyzed (Participants) | 19 | 17 | 18 | 19 | 17
participants
  TEAEs | 14 | 13 | 13 | 11 | 11
  TESAEs | 0 | 1 | 1 | 0 | 0
  Treatment related TEAEs | 3 | 4 | 2 | 2 | 3

7. Secondary Outcome: Number of Treatment-Emergent Adverse Events (TEAEs) by Severity
Description: An AE was any untoward medical occurrence attributed to study drug in a participant who received study drug. Investigator assessed TEAEs as mild (did not interfere with participant's usual function), moderate (interfered to some extent with participant's usual function) or severe (interfered significantly with participant's usual function). TEAEs are events between first dose of study drug and up to Day 141 that were absent before treatment or that worsened relative to pretreatment state.
Time Frame: Day 1 up to Day 141
Population: Safety analysis set included all participants who received at least 1 dose of study drug.
Measure: Number; unit: adverse events
Arm/Group | Placebo | PF-04950615 0.25 mg/kg | PF-04950615 1.0 mg/kg | PF-04950615 3.0 mg/kg | PF-04950615 6.0 mg/kg
Number analyzed (Participants) | 19 | 17 | 18 | 19 | 17
adverse events
  Mild | 24 | 18 | 30 | 18 | 17
  Moderate | 2 | 16 | 13 | 12 | 10
  Severe | 0 | 1 | 1 | 0 | 0

8. Secondary Outcome: Number of Participants With Clinically Relevant Laboratory Abnormalities
Description: Hematology (hemoglobin[hgb],hematocrit,red blood cell[RBC]<0.8*lower limit of normal[LLN],mean cell[MC] volume,MC hgb,MC hg concentration <0.9*LLN, greater than[>] 1.1*upper limit of normal[ULN], platelet <0.5*LLN,>1.75*ULN, white blood cell[WBC]<0.6*LLN,>1.5*ULN,neutrophil,lymphocyte <0.8*LLN,>1.2*ULN,eosinophil,basophil,monocyte >1.2*ULN);chemistry(total, direct, indirect bilirubin[BR]>1.5*ULN,aspartate aminotransferase[AT],alanine AT,alkaline phosphatase,gamma-glutyl transferase>3.0*ULN,protein,lactate dehydrogenase <0.8*LLN,>1.2*ULN,creatinine,blood urea nitrogen>1.3*ULN,uric acid >1.2*ULN,potassium,chloride,calcium,bicarbonate<0.9*LLN,>1.1*ULN, sodium<0.95*LLN,>1.05*ULN,glucose[GL]<0.6*LLN,>1.5*ULN,amylase,lipase >1.5*ULN,creatinine kinase>2.0*ULN);urinalysis(pH <4.5,>8,specific gravity<1.003 , >1.030, GL,ketone,protein,hgb,BR,nitrite,leukocyte greater than or equal to [>=]1, RBC, WBC >=20);coagulation(prothrombin[PT],PT international ratio,partial thromboplastin time>1.1*ULN).
Time Frame: Day 1 up to Day 141
Population: Safety analysis set included all participants who received at least 1 dose of study drug. Here 'N' signifies those participants who were evaluable for this outcome measure.
Measure: Number; unit: participants
Arm/Group | Placebo | PF-04950615 0.25 mg/kg | PF-04950615 1.0 mg/kg | PF-04950615 3.0 mg/kg | PF-04950615 6.0 mg/kg
Number analyzed (Participants) | 19 | 17 | 18 | 18 | 17
participants | 18 | 15 | 17 | 18 | 14

9. Secondary Outcome: Number of Participants With Clinically Significant Changes in Vital Signs and Electrocardiogram (ECG) Parameters
Description: Criteria for clinical significant vital signs: maximum increase or decrease from baseline in supine systolic blood pressure (BP) greater than or equal to (>=) 30 millimeter of mercury (mmHg), maximum increase or decrease from baseline in supine diastolic BP of >=20 mmHg. Criteria for clinically significant ECG parameters: maximum increase of >=25 percent (%) for baseline value of >200 millisecond (msec) and maximum increase of >=50% for baseline value of less than or equal to (<=) 200 msec for PR and QRS interval; maximum increase from baseline of >30 to <=60 msec and maximum increase from baseline of >60 msec for QT interval corrected using the Fridericia's formula (QTCF).
Time Frame: Day 1 up to Day 141
Population: Safety analysis set included all participants who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | Placebo | PF-04950615 0.25 mg/kg | PF-04950615 1.0 mg/kg | PF-04950615 3.0 mg/kg | PF-04950615 6.0 mg/kg
Number analyzed (Participants) | 19 | 17 | 18 | 19 | 17
participants
  Supine systolic BP: Maximum increase >=30mmHg | 2 | 4 | 3 | 3 | 0
  Supine diastolic BP: Maximum increase >=20mmHg | 2 | 2 | 2 | 2 | 0
  Supine systolic BP: Maximum decrease >=30mmHg | 1 | 3 | 0 | 2 | 3
  Supine diastolic BP: Maximum decrease >=20mmHg | 1 | 4 | 1 | 4 | 2
  PR interval: >=25/50% increase | 0 | 0 | 0 | 0 | 0
  QRS interval: >=25/50% increase | 0 | 0 | 0 | 0 | 0
  QTCF: Maximum increase >30 to <=60 msec | 1 | 3 | 3 | 1 | 2
  QTCF: Maximum increase >60 msec | 0 | 0 | 0 | 0 | 0

10. Secondary Outcome: Number of Participants With Anti-drug Antibody (ADA)
Description: Human serum ADA samples of participants who received PF-04950615 (RN316) were analyzed for the presence of anti-PF-04950615 (RN316) antibodies by using the semi quantitative enzyme-linked immunosorbent assay (ELISA). Results with titer value >=4.32 nanogram per milliliter of anti-PF-04950615 antibodies were counted as positive. Number of participants with presence of anti-PF-04950615 antibodies were reported in this outcome measure.
Time Frame: Day 1 up to Day 141
Population: Analysis set included all participants who received at least 1 dose of PF-04950615 (RN316).
Measure: Number; unit: participants
Arm/Group | PF-04950615 0.25 mg/kg | PF-04950615 1.0 mg/kg | PF-04950615 3.0 mg/kg | PF-04950615 6.0 mg/kg
Number analyzed (Participants) | 17 | 18 | 19 | 17
participants | 0 | 3 | 1 | 1

11. Other Pre Specified Outcome: Change From Baseline in Lipoprotein (a) (Lp[a]) at Day 29, 57, 71, 85, 99, 127 and 141
Description: as for outcome 1
Time Frame: Baseline, Day 29, 57, 71, 85, 99, 127, 141
Population: Efficacy analysis set. 'number analyzed' = participants who were evaluable for specified time points for each arm. Results for change at Day 85 in Lp(a) was not reported because data was not collected for Lp(a) at Day 85 due to an inadvertent omission in the protocol.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Placebo | PF-04950615 0.25 mg/kg | PF-04950615 1.0 mg/kg | PF-04950615 3.0 mg/kg | PF-04950615 6.0 mg/kg
Number analyzed (Participants) | 19 | 17 | 18 | 19 | 17
mg/dL
  Baseline | 37.46 (34.809) | 61.05 (50.109) | 63.66 (50.594) | 66.29 (79.992) | 59.73 (72.611)
  Change at Day 29: number analyzed (Participants) | 19 | 16 | 17 | 18 | 14
  Change at Day 29 | 3.30 (9.837) | 2.49 (17.630) | 2.79 (21.729) | -5.42 (17.801) | -14.08 (15.693)
  Change at Day 57: number analyzed (Participants) | 17 | 15 | 15 | 18 | 17
  Change at Day 57 | 1.50 (11.677) | -2.11 (7.274) | 0.86 (22.192) | -3.44 (19.032) | -11.70 (23.474)
  Change at Day 71: number analyzed (Participants) | 18 | 15 | 17 | 17 | 17
  Change at Day 71 | 1.27 (13.458) | -0.84 (10.351) | -9.26 (24.021) | -4.57 (16.857) | -15.45 (34.324)
  Change at Day 99: number analyzed (Participants) | 19 | 17 | 17 | 18 | 16
  Change at Day 99 | 2.22 (14.847) | 4.71 (15.625) | -1.70 (10.730) | 4.89 (24.930) | -17.52 (37.185)
  Change at Day 127: number analyzed (Participants) | 19 | 16 | 17 | 17 | 16
  Change at Day 127 | -3.25 (28.197) | 2.11 (11.218) | -0.59 (19.654) | -6.45 (37.106) | -8.11 (31.751)
  Change at Day 141: number analyzed (Participants) | 19 | 17 | 18 | 17 | 16
  Change at Day 141 | 2.48 (13.753) | -0.72 (15.353) | 0.84 (12.110) | 3.93 (14.947) | -5.52 (36.935)

12. Other Pre Specified Outcome: Percent Change From Baseline in Lipoprotein (a) (Lp[a]) at Day 29, 57, 71, 85, 99, 127 and 141
Description: as for outcome 1
Time Frame: Baseline, Day 29, 57, 71, 85, 99, 127, 141
Population: Efficacy analysis set. 'number analyzed' = participants who were evaluable for specified time points for each arm. Results for percent change at Day 85 in Lp(a) was not reported because data was not collected for Lp(a) at Day 85 due to an inadvertent omission in the protocol.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | PF-04950615 0.25 mg/kg | PF-04950615 1.0 mg/kg | PF-04950615 3.0 mg/kg | PF-04950615 6.0 mg/kg
Number analyzed (Participants) | 19 | 17 | 18 | 19 | 17
percent change
  Percent change at Day 29: number analyzed (Participants) | 19 | 16 | 17 | 18 | 14
  Percent change at Day 29 | 11.56 (25.846) | 14.10 (42.815) | 4.23 (22.161) | -21.34 (25.694) | -29.90 (22.427)
  Percent change at Day 57: number analyzed (Participants) | 17 | 15 | 15 | 18 | 17
  Percent change at Day 57 | 5.13 (20.258) | -0.02 (14.398) | 1.38 (21.771) | -10.60 (22.427) | -23.43 (27.739)
  Percent change at Day 71: number analyzed (Participants) | 18 | 15 | 17 | 17 | 17
  Percent change at Day 71 | -3.14 (27.897) | -3.43 (14.579) | -21.42 (26.676) | -18.77 (23.309) | -25.95 (29.676)
  Percent change at Day 99: number analyzed (Participants) | 19 | 17 | 17 | 18 | 16
  Percent change at Day 99 | 0.20 (23.623) | 2.66 (19.043) | -3.46 (19.600) | -6.58 (5.693) | -25.39 (22.064)
  Percent change at Day 127: number analyzed (Participants) | 19 | 16 | 17 | 17 | 16
  Percent change at Day 127 | -0.08 (42.026) | 1.84 (15.518) | -0.14 (28.160) | -11.44 (31.828) | -12.93 (27.915)
  Percent change at Day 141: number analyzed (Participants) | 19 | 17 | 18 | 17 | 16
  Percent change at Day 141 | 7.37 (28.842) | -2.41 (20.150) | -1.27 (19.554) | 0.50 (22.445) | -2.41 (31.080)

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as nonserious in another participant or one participant may have experienced both a serious and nonserious event during the study. Safety population.
Arm/Group | Placebo | PF-04950615 0.25 mg/kg | PF-04950615 1.0 mg/kg | PF-04950615 3.0 mg/kg | PF-04950615 6.0 mg/kg
Serious Adverse Events (participants affected / at risk) | 0/19 | 1/17 | 1/18 | 0/19 | 0/17
Other Adverse Events (participants affected / at risk) | 14/19 | 13/17 | 13/18 | 11/19 | 11/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=19) | PF-04950615 0.25 mg/kg (N=17) | PF-04950615 1.0 mg/kg (N=18) | PF-04950615 3.0 mg/kg (N=19) | PF-04950615 6.0 mg/kg (N=17)
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Depression (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=19) | PF-04950615 0.25 mg/kg (N=17) | PF-04950615 1.0 mg/kg (N=18) | PF-04950615 3.0 mg/kg (N=19) | PF-04950615 6.0 mg/kg (N=17)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0
Sinus arrest (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Supraventricular extrasystoles (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Ventricular extrasystoles (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Ear disorder (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Hypoaesthesia oral (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Lip dry (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 1 | 0 | 1 | 0
Polyp colorectal (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Salivary hypersecretion (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0
Axillary pain (General disorders) | 0 | 1 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 1 | 1
Influenza like illness (General disorders) | 0 | 1 | 0 | 0 | 0
Infusion site phlebitis (General disorders) | 0 | 0 | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 1 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 1 | 2 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 1 | 0
Acute sinusitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Fungal skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 2
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 1 | 1 | 1 | 1 | 0
Oral herpes (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 1 | 2 | 0 | 0
Tooth abscess (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 0 | 4 | 3 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 2 | 0
Viral infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Joint injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Muscle strain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Tooth fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1 | 0 | 0
Amylase increased (Investigations) | 0 | 0 | 1 | 0 | 0
Bilirubin conjugated increased (Investigations) | 0 | 0 | 1 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 1 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 1 | 0 | 0 | 0
Blood glucose increased (Investigations) | 0 | 0 | 1 | 0 | 0
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 1 | 0 | 0
Blood pressure decreased (Investigations) | 0 | 1 | 0 | 0 | 0
Blood pressure increased (Investigations) | 0 | 1 | 0 | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 1 | 0 | 1
Lipase increased (Investigations) | 0 | 0 | 1 | 0 | 0
Occult blood positive (Investigations) | 0 | 1 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Increased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 2 | 3
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 1 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0 | 1
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 5 | 3 | 3 | 3 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 1 | 0 | 1
Hyporeflexia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Migraine (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Paraesthesia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1
Sinus headache (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Syncope (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Hypertonic bladder (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Rhinitis seasonal (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Haematoma (Vascular disorders) | 1 | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
Due to an inadvertent omission in the protocol at Day 85, presented limitations in the assessment of treatment effect on ApoA1, ApoB and Lp(a) for Day 85.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.